CLINICAL TRIAL: NCT02663739
Title: Zenith TXD Dissection Stent Graft System Usage Results Surveillance in Japan for Treating Acute Complicated Stanford Type B Aortic Dissection
Brief Title: Zenith® TXD Post-market Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-12
Record Dates: First submitted 2016-01-22; First posted 2016-01-26 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Aortic Dissection
Keywords: Stanford type B aortic dissection; Malperfusion; Rupture; Acute disease; Endovascular procedures
MeSH Terms: conditions — Aortic Dissection; Rupture; Acute Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Aortic Dissection: Treating patients with acute complicated Stanford Type B aortic dissection with the Zenith® TXD
  Interventions: Device: Zenith® TXD

INTERVENTIONS:
Device: Zenith® TXD — Zenith® TXD Dissection Stent Graft System for treatment of patients with aortic dissection of the descending thoracic aorta

SUMMARY:
The study is a post-market surveillance study required by Japanese Regulatory Authorities as a condition of approval

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic aortic dissection, including attempted cases
* Patients with acute Stanford type B aortic dissection, including attempted cases

Exclusion Criteria:

* Stanford type A aortic dissection and/or chronic type B aortic dissection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Japan treated with TXD at investigational sites.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-03; Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Rate of major adverse events | 5 years
  Major adverse events will include death, aortic rupture, conversion to open surgical repair, spinal cord ischemia, retrograde progression of dissection, myocardial infarction, renal failure requiring dialysis, intestinal ischemia, stroke, paraplegia, and > 72 hours artificial respiratory assistance.

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Kato, MD, Study Chair — Morinomiya Hospital; Kimihiko Kichikawa, MD, Study Chair — Nara Medical University Hospital; Hideyuki Shimizu, MD, Study Chair — Keio University Hospital; Joseph Lombardi, MD, Study Chair — The Cooper Health System
Locations (27):
- Japan (27):
  - Kokura Memorial Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Minami Tohoku Hospital, Fukushima
  - Iwaki Kyoritsu Hospital, Fukushima
  - Hospital Hakodate Hokkaido, Hokkaido
  - Steel Memorial Muroran Hospital, Hokkaido
  - Hyogo Brain and Heart Center, Hyōgo
  - Mie University Hospital, Mie
  - Sendai Kousei Hospital, Miyagi
  - Shinshu University Hospital, Nagoya
  - Tenri Hospital, Nara
  - University of the Ryukyus Hospital, Okinawa
  - Morinomiya Hospital, Osaka
  - Matsubara Tokushukai Hospital, Osaka
  - Kinki University Hospital, Faculty of Medicine, Osaka
  - Oita University Hospital, Ōita
  - Saitama International Medical Center, Saitama
  - Dokkyo Medical Univercity Hospital, Tochigi
  - Saiseikai Utsunomiya Hospital, Tochigi
  - Jikei University School of Medicine, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Japanese Red Cross Musashino Hospital, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata
  - Nihonkai General Hospital, Yamagata
  - Yamaguchi Grand Medical Center, Yamaguchi